CLINICAL TRIAL: NCT03276195
Title: Studies in Patients With Rett Syndrome, Tuberous Sclerosis Complex, Neurofibromatoses, and Other Neurodevelopmental Disorders
Brief Title: Studies in Patients With Tuberous Sclerosis Complex
Status: Completed | Type: Observational
Sponsor: Translational Genomics Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: vnarayanan15-016
Record Dates: First submitted 2017-04-28; First posted 2017-09-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Neurodevelopmental Disorder; Genomics; Genetics
MeSH Terms: conditions — Tuberous Sclerosis; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participant samples for this study may include blood, urine or saliva. An optional skin biopsy may also be collected. Additional samples (such as cerebrospinal fluid, muscle biopsies, and brain tissue) can be used when they are collected as part of a clinically indicated procedure.
  Where possible, parents of a child will be enrolled to identify genetic variants (genetic modifiers). These and other biological relatives will be asked to donate blood samples and optional skin biopsy samples for study participation. If the relative is unable to donate a blood sample, a saliva sample can be collected instead.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Familial TSC and families: Individuals with familial TSC including those with a clinical diagnosis but no genetic confirmation and individuals with a genetic diagnosis
- Sporadic TSC and families: Individuals with sporadic TSC including those with a clinical diagnosis but no genetic confirmation and individuals with a genetic diagnosis

SUMMARY:
This study is aimed to carry out a systematic study to examine the effects of genetic variants (genetic modifiers) other than TSC genes on phenotypic variability in familial TSC patients (affected parent, child and unaffected siblings) and sporadic TSC.

DETAILED DESCRIPTION:
Tuberous sclerosis complex (TSC) is an autosomal dominant neurogenetic disorder, caused by heterozygous mutations in at least two different genes, TSC1, and TSC2. It is estimated to affect 1 in 6000, and demonstrates both phenotypic and genetic heterogeneity. It is characterized by a variety of symptoms including skin lesions, renal angiomyolipomas, cardiac rhabdomyomas, seizures, and cognitive delay (mental retardation, autism, and behavior problems). The severity of the disease varies widely among patients with TSC in general, and variability in phenotype is detectable within single families, where all affected individuals have the same TSC1 or TSC2 mutation. Neurocognitive phenotypes in TSC vary from profound mental retardation, intractable epilepsy, and autism, to normal cognition and only a mild behavioral phenotype. However, the basis of this phenotypic variability is not understood. There is a growing body of literature implicating genetic variation in "modifier genes" as an agent for phenotypic heterogeneity in Mendelian disorders, such as TSC. The role of genetic modifiers on disease severity has not yet studied in familial TSC and sporadic TSC. This study is aimed to carry out a systematic study to examine the effects of genetic variants other than TSC genes on phenotypic variability in familial TSC patients (affected parent, child and unaffected siblings) and sporadic TSC. The main objectives of the study are:

1. To identify new gene mutations (genetic modifiers) in TSC familial pairs and sporadic cases that account for the phenotypic variability.
2. Determination of quantitative differences in gene expression and allelic expression imbalance between mild and severe disease phenotype.
3. Establish a specimen repository of familial and sporadic TSC cohort to validate the genetic modifiers.

To identify genetic variants that differentiate disease severity using next generation sequencing (NGS) in DNA, and gene expression profile in RNA from blood to identify disease-causing heterozygous TSC(1 or 2) mutation in parent-child (P-C) pairs and sporadic cases with a mild and severe form of the disease. Use of next-generation sequencing (NGS) along with improved data analysis in this proposal will overcome many of the barriers in identifying genetic modifiers. The investigators will also study cultured fibroblasts cells and buccal swabs from P-C pairs to validate the findings. Use of next-generation sequencing (NGS) along with improved data analysis in this proposal will overcome many of the barriers in identifying genetic modifiers. This research has the potential to address a critical scientific gap in understanding the phenotypic variability The investigators may be able to develop a "molecular profile" that correlates with and predicts disease severity. The findings may provide a tool for early prediction of disease severity, allowing for the use of disease modifying treatments that may prevent the development of a severe neurocognitive phenotype.

As this is not a treatment protocol, there is no primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial TSC or sporadic TSC, or a biological relative of a person diagnosed with such a disorder.
* Willingness and ability to donate biospecimens to TGen for the purpose of propelling research. The minimum biospecimen donation capability is saliva and/or cheek swab. In most cases, blood or other tissue (skin biopsy) may be the ideal sample for study.

Exclusion Criteria:

* Individuals that are 18 years or older that lack the capacity to consent for themselves.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll subjects affected with Tuberous Sclerosis Complex (either familial or sporadic) and biological relatives (primarily the individual's parents or siblings). This study will consist of 1000 families who have an individual affected with TSC and wish to donate samples.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Next Generation Sequencing to Measure Phenotypic Variability | Up to 4 Years
  Identify genetic variants and disease mechanisms responsible for phenotypic variability among patients who are diagnosed with Tuberous Sclerosis Complex (TSC) and their family members.

CONTACTS AND LOCATIONS:
Overall Officials: Vinodh Narayanan, Principal Investigator — Translational Genomics Research Institiute (TGen)
Locations (1):
- Translational Genomics Research Institute (TGen), Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant study data will be published to a central data repository that allows qualified research scientists to access and look at the data under controlled access.
Time Frame: 6 months after completion of the study
Access Criteria: This data will be available to qualified researchers under controlled access